CLINICAL TRIAL: NCT04059146
Title: Tendinopathy Education on the Achilles
Acronym: TEAch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruth Chimenti (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ruth Chimenti, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201904722
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Results first posted 2023-01-11 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to type of education program Outcomes assessor will be blinded to treatment group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Education + Exercise (Experimental): The goals of the pain education intervention are for patients to 1) address fear of movement and pain catastrophizing specific to AT, 2) learn about the neurophysiology of pain, 3) develop coping skills, and 4) promote exercise participation through pacing. This program enables patients to have a conceptual change in their understanding of what causes pain, gain greater control over the psychological aspects of pain, and reduce the perceived threat of chronic pain.
  All participants will receive the same progressive Achilles tendon loading exercise program.
  Interventions: Other: Pain Education and Exercise
- Standard Education + Exercise (Active Comparator): The comparison group will be given education based on standard of care resources that primarily utilize a biomedical model, which assumes that AT pain is primarily caused by tissue damage.
  All participants will receive the same progressive Achilles tendon loading exercise program.
  Interventions: Other: Standard Education and Exercise

INTERVENTIONS:
Other: Pain Education and Exercise — Participants will be randomly assigned to a pain education group, following biopsychosocial model, or standard of care education, following biomedical model. The goals of the pain education intervention are for patients to 1) address fear of movement and pain catastrophizing specific to AT, 2) learn about the neurophysiology of pain, 3) develop coping skills, and 4) promote exercise participation through pacing. This program enables patients to have a conceptual change in their understanding of what causes pain, gain greater control over the psychological aspects of pain, and reduce the perceived threat of chronic pain. Participants will be given weekly online exercises to promote engagement with the material, give individual feedback to participants, and assess understanding. In person sessions with the physical therapist will reinforce self-learning and application to a home exercise program.
  Arms: Pain Education + Exercise
Other: Standard Education and Exercise — The comparison group will be given education based on standard of care resources that primarily utilize a biomedical model, which assumes that AT pain is primarily caused by tissue damage. The videos, handouts, and exercises will be equivalent to the pain education group in terms of time and learning requirements.
  Arms: Standard Education + Exercise

SUMMARY:
This is a randomized double-blind, placebo-controlled trial with individuals who have chronic Achilles tendinopathy (AT). This study investigates the effects of education on outcomes (specified in hypotheses below) related to participation in an exercise program. Participants will be randomized to one of two educational programs. All participants will receive the same exercise intervention. This study will consent and randomize 66 participants, who will complete 2 in-person evaluation sessions (baseline, 8-week follow-up), 8 treatment sessions with a physical therapist (between baseline and 8-week follow-up), and 1 online evaluation sessions (12-week follow-up).

We hypothesize that 1) a biopsychosocial approach to education will decrease pain (NPRS) and disability (PROMIS physical function) more than the standard of care for patients with AT, 2) exercise will improve all three pain mechanisms examined in this RCT (increased PPT, decreased kinesiophobia, increased number of heel raises).

DETAILED DESCRIPTION:
This feasibility randomized controlled trial was designed to address the following aims:

Specific Aim 1 examines if education on central pain mechanisms (i.e. biopsychosocial approach) compared to education on peripheral pain mechanisms (i.e. standard of care utilizing a biomedical approach) is more effective at reducing pain and disability in a pilot RCT exercise program for Achilles tendinopathy. We hypothesize that a biopsychosocial approach to education will decrease pain (NPRS) and disability (PROMIS physical function) more than the standard of care for patients with AT.

Specific Aim 2 determines which central pain mechanisms (nociplastic pain, pain psychology, motor dysfunction) are improved by an exercise program, regardless of education group. We hypothesize that exercise will improve all three central pain mechanisms (increased PPT, decreased kinesiophobia, increased number of heel raises).

A total of 66 adults with chronic Achilles tendinopathy (AT) will be enrolled (consented and randomized) in this single-site pilot randomized controlled trial (RCT). All data will be collected at a single site within an academic medical center. A pilot RCT comparing effectiveness of exercise with pain education to standard of care, i.e. exercise with biomedical education. Participants will be randomized to treatment group using a permuted block randomization scheme stratified by sex and AT type (insertional and midportion). Participants will complete up to 7 treatment sessions over an 8-week period. With an anticipated 10% dropout rate, we plan to analyze data on 30 adults with chronic AT per group.

Participants will complete 2 evaluation sessions at baseline and 8-week follow-up. Evaluation sessions will involve the following 4 types of testing.

1. Clinical exam (including ultrasound imaging)
2. Questionnaires (demographics, symptom description, and psychological) Private, identifiable information will be collected via questionnaires administered online and in-person. All data will be entered into a University of Iowa REDCap database, which is maintained by University of Iowa ITS staff.

2) Movement analysis and verbal pain rating Participants' motion and force will be captured as they walk, perform heel raises, hop, and do calf stretches within a 3-dimensional motion analysis with force plates flush with the floor. To monitor pain level throughout participation, we will have participants verbally rate their pain with each task.

3) Sensory testing (Pain pressure threshold at the hamstring and Achilles bilaterally; Conditioned pain modulation at the Achilles)

In addition, participants will complete questionnaires at 12-weeks. Participants will attend 7 treatment sessions over approximately 8 weeks. Over this time period participants will complete the following procedures

1. Questionnaires (exercise adherence, educational quizzes, symptom description) This private, identifiable information will be collected via questionnaires administered online and in-person. All data will be entered into a University of Iowa REDCap database, which is maintained by University of Iowa ITS staff.
2. Exercise participation Participants will be given exercises to do at home in between treatment sessions. Participants will receive instruction from a physical therapist prior to doing the exercise at home.
3. Education Participants will be given homework and online quizzes to do at home in between treatment sessions. The physical therapist will review the educational material with the participant at each visit.

In addition, a research team member will access the medical records of participants with Achilles tendinopathy to gain information about the participant's medical history and imaging related to Achilles tendinopathy.

The sample size was based on a power analysis for the primary outcome measures of Specific Aims 1 and 2.

Specific Aim 1: This analysis will compare the between group (biopsychosocial vs biomedical approach to education) changes in pain and disability scores from baseline to 8 weeks and to 12-week follow-up for participants with AT participating in an exercise program. Based on findings from Moseley et al. for an RCT comparing a 4-week exercise program with education on central pain mechanisms to standard of care in 49 patients with chronic low back pain, we anticipate between group differences with Cohen's d greater than or equal to 0.36 for pain (between group difference across 2 time points=0.75, SD of 1.05 on the NPRS, effect size of f=0.36) and disability (between group difference across 2 time points=1.95, SD of 2.33 on low back pain-specific measure, effect size of f=0.42). Under these assumptions, a sample size of 30 patients per group would be needed to reach 80% power for the time averaged difference between two group means in a repeated measures design with alpha equal to 0.025 (Bonferroni correction of 0.05/2 for 2 outcomes in Aim 1) to detect a between group effect size of 0.36.

Specific Aim 2: This analysis will compare the within group changes (baseline to 8-weeks and to 12 weeks) in central pain mechanisms (nociplastic pain, psychosocial factors, motor dysfunction) with an exercise intervention for participants with AT, regardless of educational group. The power analysis for this aim is based on data from 3 studies that have had a moderate to large (Cohen's d greater than or equal to 0.51) treatment effects on central pain mechanisms. A study led by Dr. Sluka previously found that massage improved PPTs 2 days after an intense exercise protocol with a large effect size (27.6%, SD=14.7%, effect size= 1.88). Cai et al. found that a 4-week cognitive behavioral therapy program reduced fear of movement by 8.1 points with a SD of 5.44 (effect size= 1.5). Based on our preliminary data from the K99 phase, there was a mean improvement of 3.4 repetitions (SD of change= 6.7) in heel rise performance after an anesthetic injection for the AT group (effect size=0.51). We used the smallest and population-specific anticipated effect size of 0.51 to calculate the sample size for Aim 2. Type I error rate of alpha equal to 0.017 (Bonferroni correction of 0.05/3 for 3 outcomes in Aim 2) will be used for this aim to adjust for the multiple comparisons. The sample size of 60 patients calculated for Aim 1 would allow us to detect an effect size of d greater than or equal to 0.43 with 80% power under these assumptions.

The normality of the continuous data will be tested by the Shapiro-Wilk test and by examining the quantile-quantile plot. Normally distributed Continuous variables will be presented as mean plus or minus SD for normally distributed data and median with interquartile ranges for non-normally distributed data. When the normality assumption is not met, transformation, such as log, will be used to complete planned parametric analyses. Type I error rate will be maintained at 0.05 by using Bonferroni adjustment for multiple comparisons. First, potential differences between group demographics at baseline will be examined univariately using two independent samples t-tests and chi-square tests, as appropriate. If differences are observed, these variables will be used as covariates in the multivariable models.

A modified intention-to-treat principle will be followed, which will include outcome data on all participants based on the group they were randomized and complete evaluation at 8 weeks. We will also compare patient characteristics of those who remained in the study to those who dropped out to determine if data at subsequent time points is consistent with missing at random.

For Aim 1 we will assess the effect of the interventions on the primary outcomes for pain (NPRS) and disability (PROMIS physical function) from baseline to 8-weeks and to 12-week follow-up using linear mixed model for repeated measures. Similarly, for Aim 2 a linear mixed model for repeated measures will assess the effect of the interventions by group on the primary outcomes for central pain mechanisms (nociplastic pain: PPT, psychosocial factors: TSK, motor control: heel raises) from baseline to 8 weeks. For Aims 1 and 2, the factors in the linear mixed model will include group and time effects. In addition, the significance of the group*time interaction term, where the group*time interaction tests if the change over time differs between groups, will also be tested. We will also assess for normality, linearity, homoscedasticity, and independence of residuals for the multiple regression models (dependent variables: pain and disability). Statistical significance will be defined by alpha greater than or equal to 0.05.

Analyses for secondary outcome measures of central sensitization, psychological factors, motor control, pain and disability for Aims 1 and 2 will be performed using the same statistical tests described above. Secondary analyses on sex will examine potential sex-based differences in both Aims 1 and 2 to inform sample size estimates for future clinical trials. The analyses described above for each aim will be expanded to explore the effect of sex as a fixed factor and examine interactions with group and time. Using the same data analysis strategy as described for sex, a secondary analysis on AT type (insertional vs. midportion) will also be assessed for Aims 1 and 2 to inform recruitment strategies for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Primary source of pain localized to Achilles tendon insertion or midportion
* Localized pain at least 3/10 in the Achilles tendon (midportion, insertion, unilateral or bilateral) during walking, heel raises, or hopping
* Pain that increases (>1 point on 11-point scale) with increasing load

Exclusion Criteria:

* Younger than 18 years of age
* Inability to read and write in English
* Achilles tendon pain for less than 3 months
* History of Achilles tendon rupture that was verified with surgical or conservative management
* History of invasive intervention (surgery, tenex) for AT on more painful side
* Non-invasive treatment (physical therapy, nitroglycerine patch, iontophoresis, injection) for AT in the past 3 months
* Diagnosed with systemic inflammatory conditions (e.g. rheumatoid arthritis, ankylosing spondylitis), endocrine disorder with complications (e.g. Uncontrolled Type I or II diabetes, Diabetic peripheral neuropathy), connective tissue disorder (e.g. Marfan's syndrome)
* Cardiovascular conditions that may be exacerbated by a 90 second submersion of hand in cold water (Raynaud's, cold contact uticaria)
* History of taking fluoroquinolones within the past 3 months
* History of corticosteroid injection to foot/ankle/leg within the past 3 months
* Foot and ankle pain primarily due to other pathology, such as posterior impingement, bursitis, paratendonitis, sural nerve injury, ankle osteoarthritis, or radicular/referred symptoms (pain, altered sensation, weakness, altered reflexes) from lumbar spine into lower extremities
* Four step square test >15 seconds

Additional exclusion criteria for online only visits:

* Unable to successfully complete virtual visits with a webcam and/or Prefer only in-person visits
* Virtual Fall risk assessment: Stay Independent score >4[56]
* Symptoms indicating need for in-person blood pressure monitoring: 1) Inconsistent use of HTN meds, and/or 2) any recent/current associated symptoms with uncontrolled HTN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Chimenti, DPT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with FAIR data principles, data will be deposited in the University of Iowa open-access institutional repository, Iowa Research Online. The repository is open access and maintained by the Libraries at the University of Iowa for the preservation and sharing of intellectual work of faculty, students and staff.
  Datasets will be accompanied with appropriate descriptive, technical, and administrative metadata to facilitate discovery and scholarly reuse, and will be assigned unique Digital Objects Identifiers (DOIs) that can be incorporated into publications and cited in the literature. Metadata will be included in the data records in the repository through readme files and structured information following the DataCite metadata schema.
  Footnotes:
  FAIR Data Principles: https://www.go-fair.org/fair-principles/ IRO: University of Iowa. (2019). Iowa Research Online. http://ir.uiowa.edu/ DataCite metadata: https://schema.datacite.org/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available to other researchers for the primary outcomes of Specific Aims 1 and 2. Results will be posted within 1 year of study completion.
Access Criteria: The URL linking to IPD will be posted within this section and available anyone with access to clinicaltrials.gov
URL: https://doi.org/10.25820/data.006166

REFERENCES:
- [Derived] Janowski AJ, Post AA, Heredia-Rizo AM, Frey-Law LA, Bayman EO, Sluka KA, Chimenti RL. Exploring biomarkers of change in movement-evoked pain in Achilles tendinopathy: A secondary analysis of a randomized controlled trial. Clin Biomech (Bristol). 2026 Jan;131:106706. doi: 10.1016/j.clinbiomech.2025.106706. Epub 2025 Nov 7. PMID 41207117
- [Derived] Post AA, Rio EK, Sluka KA, Moseley GL, Bayman EO, Hall MM, de Cesar Netto C, Wilken JM, Danielson J, Chimenti RL. Efficacy of Telehealth for Movement-Evoked Pain in People With Chronic Achilles Tendinopathy: A Noninferiority Analysis. Phys Ther. 2023 Mar 3;103(3):pzac171. doi: 10.1093/ptj/pzac171. PMID 37172125

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Education + Exercise: The comparison group will be given education based on standard of care resources that primarily utilize a biomedical model, which assumes that AT pain is primarily caused by tissue damage.
  All participants will receive the same progressive Achilles tendon loading exercise program.
  Standard Education and Exercise: The comparison group will be given education based on standard of care resources that primarily utilize a biomedical model, which assumes that AT pain is primarily caused by tissue damage. The videos, handouts, and exercises will be equivalent to the pain education group in terms of time and learning requirements.
Period: Overall Study
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Started | 33 | 33
Completed | 33 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Education + Exercise | Standard Education + Exercise | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.9) | 44.9 (16.1) | 43.4 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 27 | 29 | 56
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Pain (Aim 1)
Description: Participants will rate pain using the numeric pain rating scale (NPRS, 11-pt scale from 0 to 10 as worst pain imaginable) during 3 single limb heel raises
Time Frame: Pre-Intervention, Post-intervention (8-week follow-up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Number analyzed (Participants) | 33 | 33
units on a scale
  0-weeks | 4.9 (2.3) | 5.2 (1.9)
  8-weeks | 1.8 (1.8) | 1.5 (1.6)

2. Primary Outcome: Self-reported Function (Aim 1)
Description: Self-reported function will be assessed with the PROMIS physical function computer adaptive test, which has a mean score of 50 and standard deviation of 10 in the general population. A higher score indicates better physical function.
Time Frame: Pre-Intervention, Post-intervention (8-week follow-up, 12-week follow-up)
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Number analyzed (Participants) | 33 | 33
t-score
  0-weeks | 49.3 (7.4) | 47.3 (6.0)
  8-weeks | 51.0 (7.8) | 50.1 (6.3)
  12-weeks | 52.4 (7.8) | 51.2 (7.2)

3. Primary Outcome: Nociplastic Pain- CPM (Aim 2)
Description: Conditioned pain modulation (CPM) at the Achilles tendon will be calculated as the % change in the pain pressure threshold (PPT) with the hand in cold water (conditioning stimulus) compared to the (PPT) room temperature water.
Time Frame: Pre-Intervention, Post-intervention (8-weeks)
Measure: Mean (Standard Deviation); unit: percentage change in PPT with cold water
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Number analyzed (Participants) | 33 | 33
percentage change in PPT with cold water
  0-weeks | 24.0 (34.0) | 28.1 (28.8)
  8-weeks | 16.6 (17.4) | 13.3 (20.0)

4. Primary Outcome: Fear of Movement
Description: Tampa Scale of Kinesiophobia (TSK) rates current level of fear about movement causing pain and injury. Scores range from 17, indicating negligible fear of movement, to 68, indicating extreme fear of pain with movement.
Time Frame: Pre-Intervention, Post-intervention (8-weeks, 12-weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Number analyzed (Participants) | 33 | 33
units on a scale
  0-weeks | 37.2 (6.2) | 37.7 (5.2)
  8-weeks | 29.4 (6.5) | 32.6 (6.1)
  12-weeks | 29.8 (7.4) | 32.3 (6.1)

5. Primary Outcome: Performance-based Function: Heel Raises
Description: Plantarflexor endurance will be quantified with the maximum number of repetitions of single limb heel raises
Time Frame: Pre-Intervention, Post-intervention (8-weeks)
Measure: Mean (Standard Deviation); unit: Heel raises
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
Number analyzed (Participants) | 33 | 33
Heel raises
  0-weeks | 15.0 (8.5) | 18.1 (13.0)
  8-weeks | 22.3 (10.2) | 21.1 (10.6)

6. Other Pre Specified Outcome: Demographics
Description: date of birth, sex, race/ethnicity, height/weight/BMI, description of Achilles tendinopathy symptoms, goals for physical therapy, previous experience with conservative care, comorbidities
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Four Square Step Test
Description: Participants will perform a series of steps in a square formation. The duration of time needed to complete the step reflects dynamic balance and mobility.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected before and after at all evaluation and treatment visits (0-weeks to 12-weeks)
Arm/Group | Pain Education + Exercise | Standard Education + Exercise
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 4/33 | 7/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Education + Exercise (N=33) | Standard Education + Exercise (N=33)
Mild AE: Increased Achilles tendon pain with activity (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) — Achilles tendon discomfort that is reported at a treatment visit and doesn't resolve after activity modification. A mild AE may have none to mild impact study participation (<50% of evaluation and <50% of treatment progression affected).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04059146/Prot_SAP_000.pdf